CLINICAL TRIAL: NCT00177437
Title: Home Screening for Chlamydia Surveillance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0404024
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Chlamydia Trachomatis; Gonorrhea
MeSH Terms: conditions — Gonorrhea

INTERVENTIONS:
Behavioral: home testing kit

SUMMARY:
This is a randomized controlled trial to determine whether a home screening test for chlamydia and gonorrhea will lead to increased use of screening tests and increased detection of sexually transmitted diseases.

DETAILED DESCRIPTION:
This is a phase III randomized controlled trial. We enrolled 403 young women from a variety of clinical settings and neighborhoods in the Pittsburgh, PA region. Women completed a baseline questionnaire and then were randomized to either an intervention group (receive home testing kit every six months) or to a control group (receive a letter suggesting a clinic visit for screening). Participants were followed for 2 years, and medical chart abstraction was done to document tests done in clinical settings. The final study end points were number of tests completed, number of screening tests completed, number of STDs detected, and incident cases of pelvic inflammatory disease.

ELIGIBILITY:
Inclusion Criteria: age 15 to 29, 2 or more risk factors for STDs, sexually active -

Exclusion Criteria: currently pregnant, homeless

-

Ages: 15 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 403
Dates: Start 1999-06; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
chlamydia and gonorrhea tests completed
chlamydia and gonorrhea infections detected

SECONDARY OUTCOMES:
pelvic inflammatory disease cases detected

CONTACTS AND LOCATIONS:
Overall Officials: Roberta B Ness, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Cook RL, Ostergaard L, Hillier SL, Murray PJ, Chang CC, Comer DM, Ness RB; DAISY study team. Home screening for sexually transmitted diseases in high-risk young women: randomised controlled trial. Sex Transm Infect. 2007 Jul;83(4):286-91. doi: 10.1136/sti.2006.023762. Epub 2007 Feb 14. PMID 17301105